CLINICAL TRIAL: NCT04111562
Title: Does Cranioplasty Reduce Disability in Cases With Post Traumatic Skull Bone Defects
Acronym: Cranioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Salah Shaltout, Lecturer in forensic medicine and clinical toxicology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cranioplasty2018; Assiut University (Other: Assiut University Hospitals)
Record Dates: First submitted 2019-02-25; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cranioplasty; Disability Physical; Trauma
Keywords: Cranial defect; skull bone defects
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- polymethyl methacrylate Cranioplasty (Other): The Cranioplastic kit used (Teknimed, Biomaterials Innovation, Gentafix 1 ®, France) a biocompatible material that is composed of powder and liquid form of polymethyl methacrylate.
  Interventions: Procedure: Cranioplasty

INTERVENTIONS:
Procedure: Cranioplasty — Bone grafts

SUMMARY:
Background: The percentage of permanent infirmities following traumatic cranial bone cranial bone defects following trauma for restoration of function and cosmoses. This study designed to evaluate the influence of cranioplasty as a method of skull repair on work capability of the patients and their employability.

Methods: The authors compared the work capability and employment of 35 patients with traumatic cranial bone defects after head trauma treated in the Neurosurgery Department of Assiut University Hospitals, Egypt from January 2013 to January 2018 before and after cranioplasty.

DETAILED DESCRIPTION:
Cranioplasty is surgical repair of a cranial bone defect, important to cover defects following skull trauma for restoration of function, cosmoses and protective effects. Cranioplasty is the surgical procedure in which the autologous skull, synthetic materials (titanium, methyl methacrylate, polyetheretherketone implants, hydroxyapatite, and bioceramics are used to repair the skull defect

ELIGIBILITY:
Inclusion Criteria:

• Patients with traumatic skull bone defects

Exclusion Criteria:

• Patients were not working before trauma

Ages: 14 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2020-03-03 (Estimated); Study Completion 2020-03-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complications | 6 months up to one year
  the number of patients with complications after cranioplasty as a method of skull repair.

CONTACTS AND LOCATIONS:
Locations (1):
- Emanaalah shaltouy@yahoo.com, Asyut, Egypt